CLINICAL TRIAL: NCT01995656
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Oral Doses of LY3108743 in Healthy Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3108743 in Healthy Participants and Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15197; I7D-FW-SGAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo - Healthy (Placebo Comparator): Part A. Healthy participants will receive a single oral dose of placebo matching LY3108732 in at least 1 of 3 study periods.
  Interventions: Drug: Placebo - Capsule
- LY3108743 - Healthy (Experimental): Part A. Healthy participants will receive a single oral dose of LY3108743 in dose escalation cohorts in up to 2 of 3 study periods.
  Interventions: Drug: LY3108743 - Capsule
- Placebo - Diabetes (Placebo Comparator): Part B. Participants with diabetes mellitus will receive a single oral dose of placebo matching LY3108732 in at least 1 of 3 study periods.
  Interventions: Drug: Placebo - Capsule
- LY3108743 - Diabetes (Experimental): Part B. Participants with diabetes mellitus will receive a single oral dose of LY3108743 in dose escalation cohorts in up to 2 of 3 study periods.
  Interventions: Drug: LY3108743 - Capsule
- Placebo - Solution (Placebo Comparator): Part C. Contingent on results from Parts A and B. Healthy participants will receive a single oral dose of placebo matching LY3108743 in 1 of 2 study periods.
  Interventions: Drug: Placebo - Solution
- LY3108743 - Solution (Experimental): Part C. Contingent on results from Parts A and B. Healthy participants will receive a single oral dose of LY3108743 in 1 of 2 study periods.
  Interventions: Drug: LY3108743 - Solution

INTERVENTIONS:
Drug: Placebo - Capsule — Administered orally
  Arms: Placebo - Diabetes; Placebo - Healthy
Drug: LY3108743 - Capsule — Administered orally
  Arms: LY3108743 - Diabetes; LY3108743 - Healthy
Drug: Placebo - Solution — Administered orally
  Arms: Placebo - Solution
Drug: LY3108743 - Solution — Administered orally
  Arms: LY3108743 - Solution

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug known as LY3108743 in healthy participants and in participants with type 2 diabetes.

The study will also investigate how LY3108743 affects the levels of blood sugar and other naturally occurring substances (e.g. hormones that control the way sugar is used) in the body, how much of the study drug gets into the blood stream, and how long it takes the body to get rid of it.

Information about any side effects that may occur will be collected. The study is expected to last approximately 7 to 8 weeks for each participant.

The study will have up to 3 parts. Participants may enroll in only one part.

ELIGIBILITY:
Inclusion Criteria:

* Must be a male, or a female who cannot become pregnant, and who is either a healthy participant, or who has type 2 diabetes
* Have a body mass index (BMI) of 18.5 to 40.0 kilogram per square meter (kg/m^2), inclusive, at screening
* Have normal blood pressure
* Participants with diabetes must not be taking any anti-hyperglycemic medications with the exception of metformin. If on metformin, participants must be on a stable treatment regimen for at least for 4 weeks prior to screening
* Participants with diabetes must have a hemoglobin A1c (HbA1c) level between 6 to 11%, inclusive, at screening

Exclusion Criteria:

* Have previously completed or withdrawn from this study
* Have or used to have health problems or laboratory test results or electrocardiogram (ECG) readings that, in the opinion of the doctor, could make it unsafe to participate or could interfere with understanding the results of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Pre-dose up to Day 6 (5 days post-dose)

SECONDARY OUTCOMES:
Maximum Change from Baseline up to 24 Hours in Level of Blood Glucose Before and After a Standard Meal | Baseline up to 24 hours
Pharmacokinetics: Maximum Concentration (Cmax) of LY3108743 | Baseline up to 48 hours
Pharmacokinetics: Area Under the Curve (AUC) of LY3108743 | Baseline up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore